CLINICAL TRIAL: NCT04567212
Title: Gender Differences and SNPs in Asthmatic Patients
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Catanzaro (Other)
Collaborators: Azienda Sanitaria Provinciale Di Catanzaro (Other); Azienda Ospedaliera Universitaria Mater Domini, Catanzaro (Other)
Responsible Party: Principal Investigator, Luca Gallelli, MD PhD, University of Catanzaro
Other Study IDs: SNPS asthma
Record Dates: First submitted 2020-09-11; First posted 2020-09-28 (Actual); Last update posted 2020-11-23 (Actual); Status verified 2020-11

CONDITIONS: Allergic Asthma; Asthma
Keywords: asthma; allergy; Gender; polymorphism
MeSH Terms: conditions — Asthma; Hypersensitivity; Coitus

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — we will take the oral swab in order to evaluate the enzyme expression
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male-group: in this group we will enroll only male with asthma
  Interventions: Genetic: genetic evaluation; Other: MicroRNA evaluation
- Female-group: in this group we will enroll only female with asthma
  Interventions: Genetic: genetic evaluation; Other: MicroRNA evaluation

INTERVENTIONS:
Genetic: genetic evaluation — A sampe of blood (3 mL) and of oral mucosa will be take and analyzed using nCounter GX Human Inflammation Kit a comprehensive number of 8SNPs in 3 human genes known to be differentially expressed in allergic asthma.
Other: MicroRNA evaluation — Using the sampe of blood (3 mL) using RT-PCR we will evaluate the expression of microRNA in enrolled patients

SUMMARY:
The GINA 2020 guidelines suggest that asthma affects approximately 300 million persons worldwide. Even if there is a specific drug treatment for each stage of disease (From mild to severe) in some patients it is not efficacy and it culd be reated to the gender difference Polymorphisms seems to be involved in asthma (allergic or not) even if no data have been published concerning the role of gender in this clinical manifestation. The aim of this study is to assess whether genetic variations involved in the genes encoding the two key leukotriene enzymes, ALOX5 and LTC4S, and CysLTR1 are implicated in the sex difference of allergic asthma in a well-characterized patient cohort.

DETAILED DESCRIPTION:
The GINA 2020 guidelines suggest that asthma affects approximately 300 million persons worldwide. Even if there is a specific drug treatment for each stage of disease (From mild to severe) in some patients it is not efficacy and it culd be reated to the gender difference Polymorphisms seems to be involved in asthma (allergic or not) even if no data have been published concerning the role of gender in this clinical manifestation. The role of polymorphisms in susceptibility to allergic asthma has been partially investigated but no study has analysed gender subgroups separately, neglecting a their potential predictive role in symptomatological and functional variations in the allergic asthma in both sexes. The aim of this study is to assess whether genetic variations involved in the genes encoding the two key leukotriene enzymes, ALOX5 and LTC4S, and CysLTR1 are implicated in the sex difference of allergic asthma in a well-characterized patient cohort.

ELIGIBILITY:
Inclusion Criteria:

* asthma (allergic or not) diagnosed according to Global Initiative for Asthma guidelines (GINA 2020).
* signed informed consent

Exclusion Criteria:

* • infectious diseases

  * neurodegenerative diseases
  * autoimmune diseases
  * neoplasms
  * progressive serious medical conditions (such as cancer, AIDS or end-stage renal disease)
  * alcohol consumption (>3 alcoholic beverages daily)
  * substanceabuse
  * inability to give written informed consent
  * those who will not sign the consent to the processing of personal data

Ages: 6 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We will perform an observational study in patients with asthma enrolled fro general practitioners and specialist in respiratory disease. After the recruitment a sample of blood and oral mucosa will be taken to evaluate the expression of SNPs and of inflammatory status
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-08-01 (Actual); Primary Completion 2021-11-20 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Expression of SNPs | 1 month
  statistically significant difference (P<0.05) in SNPs expression between male and female

SECONDARY OUTCOMES:
Concentration of MicroRNA | 1 month
  statistically significant difference (P<0.05) in microRNA between male and female
SNPs and age | 1 month
  statistically significant difference (P<0.05) in SNPs expression between age > 12 years and < 12 years

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - AO Materdomini, Catanzaro, Italia
  - ASP Catanzaro, Catanzaro

IPD SHARING:
Plan to Share IPD: No